CLINICAL TRIAL: NCT04251143
Title: Dresden Corneal Disease and Treatment Study - Analysis for Quality Inspection of Follow-up and Treatment Procedures of Corneal Diseases of the Department of Ophthalmology (University Hospital Carl Gustav Carus Dresden)
Brief Title: Dresden Corneal Disease and Treatment Study
Status: Recruiting | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Other Study IDs: EK 104032018
Record Dates: First submitted 2020-01-30; First posted 2020-01-31 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Corneal Ectasia; Corneal Disease; Corneal Astigmatism; Keratoconus; Keratopathy
Keywords: Cornea; Ectasia; Keratoconus; Cross-Linking; Keratoplasty
MeSH Terms: conditions — Corneal Diseases; Astigmatism; Keratoconus; Dilatation, Pathologic | interventions — Corneal Cross-Linking; Corneal Topography; Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Ectasia: Keratoconus, Keratoconus suspects
  Interventions: Procedure: corneal cross-linking; Diagnostic Test: corneal topography and tomography

INTERVENTIONS:
Procedure: corneal cross-linking — UV-A Irradiation and riboflavin
Diagnostic Test: corneal topography and tomography — Detailed Information about corneal tomography is used for diagnosis

SUMMARY:
The purpose of this study is long-term follow up of patients with corneal diseases to analyze the quality of surgical interventions and diagnosis. Corneal ectasia, especially keratoconus, is a corneal disease that leads to an irreversible loss of visual acuity while the cornea becomes steeper, thinner and irregular. For these patients, surgical intervention (e.g. corneal cross-linking) is performed, in case of disease progression. Overall, a long-term follow up is needed to evaluate an early disease progression as well as corneal stability after surgical intervention.

DETAILED DESCRIPTION:
Corneal ectasia (e.g. keratoconus) is a corneal disease that is characterized by irregular steepening of corneal curvature, stromal thinning and reduced biomechanical properties. As a result of this, visual acuity is reduced and can improved by spectacles in early state or with rigid gas permeable contact lenses in mild as well as advanced stage of the disease. Furthermore, in moderate and advanced cases stromal scarring occurs that affected the vision negatively. Therefore, a corneal transplantation is needed. Since the introduction of corneal cross-linking, the amount of corneal transplantations has been reduced. It is necessary to perform closely examinations to detect the progression of the disease as well as post-operatively follow-ups to confirm treatment success.

Parameters being analyzed are:

Age, sex, refraction, family history, known duration of ectasia, previous ocular surgery, systemic diseases, systemic and topical medication;

biomicroscopy, anterior optical coherence tomography (OCT), Scheimpflug-based tomography (Pentacam), Biomechanical assessment (Ocular Response Analyzer and Corneal Visualization with the Scheimpflug Technology), optical biometry, confocal microscopy, endothelium cell count.

ELIGIBILITY:
Inclusion Criteria:

* corneal disease
* corneal ectasia

Exclusion Criteria:

* pregnancy
* age under 18 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with corneal diseases attending a University Hospital Corneal Diseases Service.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2018-03-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Follow-up intervals | 15 years
  To find the best follow-up intervals for keratoconus patients with or without progression of the disease
postoperative follow-up intervals | 15 years
  To find the best follow-up intervals for keratoconus patients after surgical Intervention.

SECONDARY OUTCOMES:
Assessment of treatment quality | 15 years
  What is the best treatment option for the individual patient?

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Raiskup, MD, PhD, Study Director — Department of Ophthalmology; Medical Faculty Carl Gustav Carus, Techinal University Dresden
Locations (1):
- Department of Ophthalmology; Medical Faculty Carl Gustav Carus; Technical University Dresden, Dresden, Saxony, Germany

REFERENCES:
- [Derived] Herber R, Lenk J, Pillunat LE, Raiskup F. Comparison of corneal tomography using a novel swept-source optical coherence tomographer and rotating Scheimpflug system in normal and keratoconus eyes: repeatability and agreement analysis. Eye Vis (Lond). 2022 May 23;9(1):19. doi: 10.1186/s40662-022-00290-6. PMID 35606839
- [Derived] Herber R, Pillunat LE, Raiskup F. Development of a classification system based on corneal biomechanical properties using artificial intelligence predicting keratoconus severity. Eye Vis (Lond). 2021 Jun 1;8(1):21. doi: 10.1186/s40662-021-00244-4. PMID 34059127